CLINICAL TRIAL: NCT02647008
Title: Pain Relief During Unsedated Office Hysteroscopy by Applying Transcutaneous Electrical Nerve Stimulation (TENS): A Randomized Double-blind Placebo-controlled Trial
Brief Title: Pain Relief During Unsedated Office Hysteroscopy by Applying TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-2
Record Dates: First submitted 2016-01-03; First posted 2016-01-06 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Uterus Dysfunction
Keywords: outpatient hysteroscopy, TENS
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ACTIVE TENS (Experimental): ACTIVE TENS
  Interventions: Device: TENS
- PLACEBO (Placebo Comparator): INACTIVE TENS
  Interventions: Device: TENS
- CONTROL (No Intervention): NO TENS

INTERVENTIONS:
Device: TENS — Transcutaneous electrical nerve stimulation (TENS) is a nonpharmacological intervention that activates a complex neuronal network to reduce pain by activating descending inhibitory systems in the central nervous system to reduce hyperalgesia.These small battery powered devices deliver alternating current via cutaneous electrodes positioned near the painful area.
  Arms: ACTIVE TENS; PLACEBO

SUMMARY:
Aim: To compare the pain-relieving effect of a specific application of TENS vs. placebo TENS and a control group during unsedated diagnostic office hysteroscopy.

Design: double-blind randomized placebo-controlled trial. Setting: Outpatient setting. Population: Women who attended annual gynecological check up, and were indicated for diagnostic office hysteroscopy.

DETAILED DESCRIPTION:
Nowadays, diagnostic hysteroscopy is an easy and economically acceptable technique, that is being used by the gynecologist to evaluate different pathologies that used to be studied by other blind techniques. Although most women tolerate it well, the most common cause for failure during office hysteroscopy is pain. In order to overcome this adversity several studies have been carried out using different types of pain relievers as local anesthesia, misoprostol, music, and NSAID to prevent the occurrence of a vagal reaction, but the results have been contradictory. Other analgesic alternatives that prioritize these three points should be considered. Transcutaneous electrical nerve stimulation (TENS) has become a very common electrotherapy as a pain-reliever because of its attributes, namely a noninvasive and non-pharmacological method based on the delivery of pulsed electrical currents through the skin, using surface electrodes, effective in many variety of conditions, such as neuropathic pain, musculoskeletal pain, headache, gynecological and obstetric pain, to treat both chronic and acute pain, even from visceral organs.

Aim: to compare the pain-relieving effect of a specific application of TENS vs. placebo TENS and a control group during unsedated diagnostic office hysteroscopy.

Design: double-blind randomized placebo-controlled trial. Setting: Outpatient setting; Hospital Provincial de Castellon (Spain) and Hospital General de Castellon (Spain).

Population: Women who attended annual gynecological check up, and were indicated for diagnostic office hysteroscopy

ELIGIBILITY:
Inclusion Criteria: women who attended annual gynecological check up, and were indicated for diagnostic office hysteroscopy because of different pathologies such as:

* postmenopausal endometrial thickening >4mm;
* postmenopausal abnormal uterine bleeding;
* suspicious endometrial polyp or leiomyoma;
* infertility study;
* suspicious endometrial carcinoma;
* hypermenorrhea

Exclusion Criteria:

* age less than 18;
* previous cervical surgery;
* neurological deficit;
* chronic or preprocedural use of opioids or psychoactive drugs;
* previous experience in TENS;
* cutaneous damage on the application sites;
* pacemakers or automatic implanted cardiac defibrillators;
* refusal to sign the informed consent form;
* inability to understand informed consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pain, assessed by visual analogue scale (VAS) | 5 minutes after hysteroscopy

SECONDARY OUTCOMES:
Pain assessed by Likert scale. | 5 minutes after hysteroscopy

OTHER OUTCOMES:
Heart Rate | 5 minutes after hysteroscopy
Blood Pleasure | 5 minutes after hysteroscopy
Total procedure time | 5 minutes after hysteroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Juan Fco. Lisón, Dr, Principal Investigator — University CEU Cardenal Herrera
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amer-Cuenca JJ, Goicoechea C, Girona-Lopez A, Andreu-Plaza JL, Palao-Roman R, Martinez-Santa G, Lison JF. Pain relief by applying transcutaneous electrical nerve stimulation (TENS) during unsedated colonoscopy: a randomized double-blind placebo-controlled trial. Eur J Pain. 2011 Jan;15(1):29-35. doi: 10.1016/j.ejpain.2010.05.006. Epub 2010 Jun 9. PMID 20538494
- [Derived] Lison JF, Amer-Cuenca JJ, Piquer-Marti S, Benavent-Caballer V, Bivia-Roig G, Marin-Buck A. Transcutaneous Nerve Stimulation for Pain Relief During Office Hysteroscopy: A Randomized Controlled Trial. Obstet Gynecol. 2017 Feb;129(2):363-370. doi: 10.1097/AOG.0000000000001842. PMID 28079781